CLINICAL TRIAL: NCT05029505
Title: Patellar Stabilization Surgery: Can the Caton-Deschamps Index be Useful in Planning?
Brief Title: The Caton-Deschamps Index Reliability in Patellar Stabilization Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: CATON
Record Dates: First submitted 2021-07-17; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Patellar Instability
Keywords: Patello-femoral Joint; Caton Deschamps Index; Patellar instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recurrent patellofemoral instability is a multifactorial pathology based on limb alignment, soft tissue constraints as well as patella and trochlear groove abnormal anatomy. For a correct and effective surgical approach, an accurate radiological evaluation is essential, which consists of the evaluation of three main factors of instability: trochlear dysplasia, abnormal height of the patella and pathological distance of the anterior tibial apophysis and trochlear throat (TA-GT). Concerning patellar height, one of the most used methods is the calculation of the Caton-Deschamps radiographic index. However, to date there is no study that certifies its reproducibility and reliability from a pre-operative assessment and planning perspective.

DETAILED DESCRIPTION:
The patellofemoral joint (PFJ) consists of two bony components, the patella and the femoral trochlea, sharing the same joint surface (1). It may be prone to instability, that is when the patella dislocates, usually on the lateral side of the knee. The incidence of primary patellar dislocation has been reported to be 5.8 cases per 100,000 in the general population, with the highest incidence occurring in the 2nd decade of life (29 per 100,000) (2). Patellar instability can be classified as traumatic, when the dislocation is caused by an external force, or nontraumatic, when native anatomy of the knee predisposes to instability. Non-operative treatment is usually taken into account for first episode of lateral patellar dislocation, unless the presence of loose bodies is verified, and consists of knee immobilization, physical therapy, non-steroidal anti-inflammatory drugs (NSAIDs) administration (3). Recurrence rate after conservative management can be up to 15-44% and patients with a clinical history of two or more dislocations have a 50% chance of recurrent dislocation episodes (4). Recurrent instability is a multifactorial problem that rely on limb alignment, bone anatomy of the patella and the trochlear groove, soft-tissue constraints, especially the medial patello-femoral ligament (MPFL). The management of recurrent patellar instability is difficult for many reasons, including heterogeneous patient population, skeletal maturity, challenging surgical approach and lack of long-term and robust clinical outcome studies (5,6). Radiologic evaluation should study the three principal factors of instability: trochlear dysplasia, abnormal patellar height, pathological tibial tubercle-trochlear groove (TT-TG) distance (7). Patellar height can be easily assessed, through standard lateral view radiographs. Several indexes for studying and calculating patellar height have been described in the literature (8-10). In patellar instability, the use of Caton-Deschamps index CDI to measure patellar height one of the most employed. Specifically, CDI relies upon the length of the articular surface of the patella and its distance from the tibia. The purpose of our study is to evaluate the reliability and reproducibility of CDI in measuring patellar height for planning patella stabilization surgery. The secondary target is to hypothesize a quantitative method of preoperative planning for anterior tibial apophysis transposition surgery, by calculating CDI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent patellar instability (≥ 2 episodes) at the time of surgery
* Indications for patellar stabilization surgery
* Availability of X-rays in digital format
* Patients who do not meet the inclusion criteria

Exclusion Criteria:

* Clinical history of <2 patella dislocations
* Non-availability of X-rays in digital format
* Not indicated for patellar stabilization surgery
* Contraindications to surgery
* Patients with osteoarthritis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from recurrent patellar instability (≥ 2 episodes) with indication of patellar stabilization surgery by reconstruction of the medial patellofemoral ligament and / or transposition of the anterior tibial tuberosity.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Caton-Deschamps index reproducibility | 6 months
  Evaluation of the Caton-Deschamps index's reproducibility in the measurement of patellar height for planning the intervention to stabilize the patella.

SECONDARY OUTCOMES:
Caton-Deschamps index reliability | 6 months
  To evaluate the reliability of the Caton-Deschamps index in measuring the patellar height for planning the intervention to stabilize the patella
Pre-operative planning | 6 months
  To hypothesize a quantitative method of preoperative planning that allows, using a mathematical calculation, to establish the extent of lowering of the patella in millimeters necessary to obtain a normal value of the Caton-Deschamps index, using radiographs with a reference calibrated at twenty millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Elisa G Pandini, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi; Roberto D'Anchise, MD, Study Director — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy